CLINICAL TRIAL: NCT07340177
Title: An Open-label, Multicenter, Randomized Controlled Clinical Trial of Xiaojin Pill/Neixiao Luoli Pill for the Treatment of Thyroid Nodules
Brief Title: Xiaojin Pill/Neixiao Luoli Pill for the Treatment of Thyroid Nodules
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, zhengchuanming, Principal Investigator, Zhejiang Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2025175
Record Dates: First submitted 2025-12-20; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Thyroid Nodules
Keywords: Thyroid nodule
MeSH Terms: conditions — Thyroid Nodule | interventions — xiaojin wan

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lifestyle Intervention + Xiaojin Pill (Experimental): Participants receive lifestyle intervention combined with oral Xiaojin Pill for the management of thyroid nodules.
  Interventions: Drug: Xiaojin Pill; Behavioral: Lifestyle Intervention
- Lifestyle Intervention + Neixiao Luoli Pill (Experimental): Participants receive lifestyle intervention combined with oral Neixiao Luoli Pill for the management of thyroid nodules.
  Interventions: Drug: Neixiao Luoli Pill; Behavioral: Lifestyle Intervention
- Lifestyle Intervention Alone (Active Comparator): Participants receive lifestyle intervention alone without study medication.
  Interventions: Behavioral: Lifestyle Intervention

INTERVENTIONS:
Drug: Xiaojin Pill — Xiaojin Pill is a traditional Chinese patent medicine administered orally at a dose of 3 g twice daily for 12 weeks.
  Other Names: Xiaojin Wan
  Arms: Lifestyle Intervention + Xiaojin Pill
Drug: Neixiao Luoli Pill — Neixiao Luoli Pill is a traditional Chinese patent medicine administered orally at a dose of 9 g twice daily for 12 weeks.
  Other Names: Neixiao Luoli Wan
  Arms: Lifestyle Intervention + Neixiao Luoli Pill
Behavioral: Lifestyle Intervention — Lifestyle intervention includes stress management, emotional regulation, healthy diet, balanced iodine intake, avoidance of smoking and alcohol, adequate rest, and reduction of radiation exposure.

SUMMARY:
The goal of this clinical trial is to learn whether Xiaojin Pill or Neixiao Luoli Pill can safely treat thyroid nodules in adults aged 18 to 65 years with benign or low-risk thyroid nodules. The main questions it aims to answer are:

* Does treatment with Xiaojin Pill or Neixiao Luoli Pill lower the size of thyroid nodules compared with lifestyle intervention alone?
* Do Xiaojin Pill or Neixiao Luoli Pill improve thyroid nodule-related symptoms and ultrasound findings while remaining safe to use?

Researchers will compare lifestyle intervention plus Xiaojin Pill, lifestyle intervention plus Neixiao Luoli Pill, and lifestyle intervention alone to see if adding Xiaojin Pill or Neixiao Luoli Pill works better than lifestyle intervention by itself.

Participants will:

* Be randomly assigned to one of the three study groups;
* Receive lifestyle intervention guidance throughout the study;
* Take Xiaojin Pill, Neixiao Luoli Pill, or no study medicine for 12 weeks, depending on their group;
* Attend follow-up visits that include thyroid ultrasound exams, blood tests to check thyroid function and safety, and symptom assessments.

DETAILED DESCRIPTION:
This study is designed to evaluate the clinical value of adding traditional Chinese medicine to standard lifestyle intervention for the management of benign or low-risk thyroid nodules.

The trial adopts a randomized, parallel-group design conducted across multiple clinical centers. After screening and baseline assessments, eligible participants are allocated to one of three management strategies: lifestyle intervention alone or lifestyle intervention combined with one of two commonly used traditional Chinese patent medicines. The study is conducted in an open-label manner, reflecting real-world clinical practice.

All participants receive standardized lifestyle guidance throughout the study period. Participants assigned to the intervention groups additionally receive oral herbal medication for a fixed treatment duration. Clinical assessments are performed at predefined time points to monitor structural changes of thyroid nodules, functional status of the thyroid gland, symptom evolution, and treatment safety.

Thyroid ultrasound examinations are performed using standardized measurement procedures to ensure consistency across centers. Safety is continuously monitored through clinical evaluation and routine laboratory testing during the treatment and follow-up periods.

The results of this study are expected to provide evidence regarding the role of traditional Chinese medicine as an adjunct to lifestyle management in patients with thyroid nodules under active surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years.
* Diagnosed with single or multiple thyroid nodules confirmed by high-resolution ultrasound, with at least one measurable nodule.
* Thyroid nodules meeting one of the following criteria:
* ACR TI-RADS category 3 with a maximum nodule diameter ≥ 1.0 cm; or
* ACR TI-RADS category 4 or 5 nodules evaluated by fine-needle aspiration and assessed as low-risk papillary thyroid carcinoma, suitable for active surveillance, with patient consent.
* Normal thyroid function at baseline, defined as thyroid-stimulating hormone (TSH), free triiodothyronine (FT3), and free thyroxine (FT4) within the reference range.
* Traditional Chinese medicine (TCM) syndrome differentiation consistent with liver qi stagnation, blood stasis, or phlegm-dampness syndrome.
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Thyroid nodules confirmed as malignant or follicular neoplasms requiring surgical intervention, or assessed by the investigator as unsuitable for active surveillance.
* Presence of hyperthyroidism or hypothyroidism, defined as abnormal TSH, FT3, or FT4 levels.
* History of severe cardiovascular, hepatic, renal, hematologic, psychiatric, autoimmune diseases, or other malignancies.
* Pregnant or breastfeeding women, or women planning pregnancy during the study period.
* Known allergy or hypersensitivity to Xiaojin Pill, Neixiao Luoli Pill, placebo components, or any ingredients of the study medications.
* Receipt of thyroid-related surgery, radiofrequency ablation, laser ablation, radioactive iodine therapy, or other treatments that may affect thyroid nodules within 3 months prior to enrollment.
* Current use of medications known to affect thyroid function or thyroid nodules, such as amiodarone or lithium.
* Poor treatment compliance or inability to complete follow-up as judged by the investigator.
* Participation in another clinical trial during the study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Percentage Change in Thyroid Nodule Volume | Baseline and Week 12

SECONDARY OUTCOMES:
Change in Thyroid Nodule-Related Symptom Score Assessed by Visual Analog Scale (VAS) | Baseline and Week 12
  Thyroid nodule-related symptoms include neck discomfort, swallowing difficulty, pressure sensation, and voice changes, assessed using a visual analog scale (VAS), with higher scores indicating more severe symptoms.
Change in Number of Thyroid Nodules | Baseline and Week 12
Change in Thyroid Nodule Ultrasound Characteristics Assessed by Standardized Ultrasound Examination | Baseline and Week 12
  Thyroid nodule ultrasound characteristics include nodule shape, margin, echogenicity, calcification, and intranodular vascularity, assessed using standardized thyroid ultrasound examination.
Change in Thyroid Function Tests (Serum TSH, FT3, and FT4) | Baseline and Week 12
  Thyroid function is assessed by measuring serum levels of thyroid-stimulating hormone (TSH), free triiodothyronine (FT3), and free thyroxine (FT4).
Number of Participants with Adverse Events | Baseline through Week 12
  Adverse events are recorded throughout the study period and include all unfavorable medical occurrences, regardless of their relationship to the study interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Chuanming Zheng, Principal Investigator — Zhejiang Provincial People's Hospital; Yuqun Zeng, Study Chair — zhejiang provincial People's Hospitial
Locations (1):
- Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No